CLINICAL TRIAL: NCT02156323
Title: A SINGLE-CENTER, OPEN-LABEL, RANDOMIZED, TWO SEQUENCE, 3-WAY CROSSOVER STUDY TO INVESTIGATE THE INTERACTION BETWEEN MULTIPLE DOSES OF COLISTIN METHANESULFONATE SODIUM (CMS) AND MULTIPLE DOSES OF RO7033877 IN HEALTHY SUBJECTS
Brief Title: A Phase 1 Clinical Study in Healthy Volunteers to Investigate the Drug-drug Interaction Between Multiple Doses of RO7033877 and Multiple Doses of Colistin Methanesulfonate Sodium (CMS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NP29333; 2014-000108-86 (EudraCT Number)
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — CD2-associated protein

ARMS (2):
- Treatment Sequence 1 (Experimental): Participants will be randomized to one of two treatment sequences. Sequence 1 is: Period 1, RO7033877; Period 2, CMS; Period 3, RO7033877 + CMS. Each period is separated by a wash-out period of at least 6 days between last dose and start of next treatment.
  Interventions: Drug: CMS; Drug: RO7033877; Drug: RO7033877 + CMS
- Treatment Sequence 2 (Experimental): Participants will be randomized to one of two treatment sequences. Sequence 2 is: Period 1, CMS; Period 2, RO7033877; Period 3, RO7033877 + CMS. Each period is separated by a wash-out period of at least 6 days between last dose and start of next treatment.
  Interventions: Drug: CMS; Drug: RO7033877; Drug: RO7033877 + CMS

INTERVENTIONS:
Drug: CMS — Multiple doses of CMS over 2.5 days
Drug: RO7033877 — Multiple doses of RO7033877 over 2.5 days
Drug: RO7033877 + CMS — Multiple doses of RO7033877 and CMS over 2.5 days

SUMMARY:
This single center, open-label, randomized study will investigate the drug-drug interaction potential between multiple doses of RO7033877 and multiple doses of colistin methanesulfonate sodium (CMS).

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (of non childbearing potential) healthy volunteers between 18 to 55 years
* Body mass index (BMI) between 18 and 30 kg/m2
* Non smokers
* Use adequate contraception methods

Exclusion Criteria:

* Evidence of active of chronic disease
* Regular consumption of drugs of abuse
* Infection with human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV)
* History of significant allergic reactions
* Abnormal blood pressure
* Clinically significant abnormalities (e.g. cardiovascular, laboratory values)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Multiple dose pharmacokinetics of RO7033877 and colistin/CMS (as appropriate): Cmax and area under the concentration-time curve (AUC) | up to 4 days (for each period)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands